CLINICAL TRIAL: NCT02422173
Title: Effects of Different Montages of Transcranial Direct Current Stimulation on the Risk of Falls and Lower Limb Function for Acute Stroke Patients: a Randomized Controlled Trial
Brief Title: Transcranial Direct Current Stimulation on the Risk of Falls and Lower Limb Function for Acute Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Professor, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tdcs002
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Anodal tDCS (Experimental): Participants in the acute post-stroke stage will receive anodal transcranial direct current stimulation
  Interventions: Device: Anodal transcranial direct current stimulation
- Cathodal tDCS (Experimental): Participants in the acute post-stroke stage will receive cathodal transcranial direct current stimulation
  Interventions: Device: Cathodal transcranial direct current stimulation
- Bilateral tDCS (Experimental): Participants in the acute post-stroke stage will receive bilateral transcranial direct current stimulation
  Interventions: Device: Bilateral transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Participants in the acute post-stroke stage will receive sham transcranial direct current stimulation
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation — The active electrode is placed on the affected hemisphere
  Arms: Anodal tDCS
Device: Cathodal transcranial direct current stimulation — The active electrode is placed on the unaffected hemisphere
  Arms: Cathodal tDCS
Device: Bilateral transcranial direct current stimulation — The cathode and anode is positioned as active electrodes on the unaffected and affected hemisphere,respectively.
  Arms: Bilateral tDCS
Device: Sham transcranial direct current stimulation — Placebo stimulation, with emission current by only 30 seconds
  Arms: Sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) has shown promising results in the modulation of cortical excitability and the promotion of neuronal plasticity after stroke. The purpose of this study was to compare the effectiveness of three different montages of tDCS (anodal, cathodal and bilateral) in reducing the risk of falls and recovery of lower limb function in acute stroke patients.

DETAILED DESCRIPTION:
This is a randomized sham-controlled trial reported following the 2010 CONSORT guidelines. The subjects were randomly allocated into 1 of 4 groups in a double-blinded parallel study design. Each patient received 10 sessions (5 consecutive days for 2 weeks) of real or sham stimulation at 2 mA intensity and current density equivalent to 0.05 A/m2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute stroke
* Able to walk 10m independently
* High risk of falling

Exclusion Criteria:

* Severe functional limitations
* Cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Four Square Step Test | Change from Baseline in Risk of Falls at 3 months

SECONDARY OUTCOMES:
Occurrence of Falling Index | Baseline, Week 2, Week 4 and Week 12
Overall Stability Index | Baseline, Week 2, Week 4 and Week 12
Falls Efficacy Scale - International | Baseline, Week 2, Week 4 and Week 12
Berg Balance Scale | Baseline, Week 2, Week 4 and Week 12
Six-minute walk test | Baseline, Week 2, Week 4 and Week 12
Sit to Stand Test | Baseline, Week 2, Week 4 and Week 12

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411